CLINICAL TRIAL: NCT02421939
Title: A Phase 3 Open-Label, Multicenter, Randomized Study of ASP2215 Versus Salvage Chemotherapy in Patients With Relapsed or Refractory Acute Myeloid Leukemia (AML) With FLT3 Mutation
Brief Title: A Study of ASP2215 Versus Salvage Chemotherapy in Patients With Relapsed or Refractory Acute Myeloid Leukemia (AML) With FMS-like Tyrosine Kinase (FLT3) Mutation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2215-CL-0301; 2015-000140-42 (EudraCT Number)
Expanded Access: NCT03070093 (Approved for marketing)
Record Dates: First submitted 2015-04-16; First posted 2015-04-21 (Estimated); Results first posted 2019-10-17 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Leukemia, Acute Myeloid (AML)
Keywords: ASP2215; Relapsed Acute Myeloid Leukemia; FLT3 Mutation; gilteritinib; Refractory Acute Myeloid Leukemia; Acute Myeloid Leukemia (AML); XOSPATA®
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — gilteritinib; Cytarabine; Azacitidine; Mitoxantrone; Etoposide; Granulocyte Colony-Stimulating Factor; fludarabine; Idarubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Gilteritinib (Experimental): Participants received 120 mg dose (3 tablets of 40 mg) orally once a day in continuous 28-day cycles, at least 2 hours after or 1 hour before food. Gilteritinib treatment continued until participants met one of the treatment discontinuation criteria.
  Interventions: Drug: gilteritinib
- Salvage Chemotherapy (Active Comparator): Participants received chemotherapy in 28-day cycles. Participants on Low-Dose Cytarabine (LoDAC) received 20 mg of cytarabine twice daily by subcutaneous (SC) or intravenous (IV) injection for 10 days. Participants on azacitidine received 75 mg/m^2 daily by SC or IV injection for 7 days. Participants on LoDAC or azacitidine treatment continued until they met discontinuation criteria. Participants on MEC chemotherapy received mitoxantrone 8 mg/m^2 daily by IV for 5 days, etoposide 100 mg/m^2 daily by IV for 5 days and cytarabine 1000 mg/m^2 daily by IV for 5 days (days 1-5). Participants on FLAG-IDA chemotherapy received G-CSF 300 μg/m^2 daily by SC/IV for 5 days (days 1-5), fludarabine 30 mg/m^2 daily by IV for 5 days (days 2-6), cytarabine 2000 mg/m^2 daily by IV for 5 days (days 2-6) and idarubicin 10 mg/m^2 daily by IV for 3 days (days 2-4). Participants receiving MEC or FLAG-IDA received 1 cycle of therapy and were assessed for response on or after day 15.
  Interventions: Drug: LoDAC (Low Dose Cytarabine); Drug: Azacitidine; Drug: MEC (Mitoxantrone, Etoposide, Cytarabine); Drug: FLAG-IDA (Granulocyte-Colony Stimulating Factor (G-CSF), Fludarabine, Cytarabine, Idarubicin)

INTERVENTIONS:
Drug: gilteritinib — tablet, oral
  Other Names: ASP2215; XOSPATA®
  Arms: Gilteritinib
Drug: LoDAC (Low Dose Cytarabine) — subcutaneous (SC) or intravenous (IV) injection
  Arms: Salvage Chemotherapy
Drug: Azacitidine — SC or IV injection
  Arms: Salvage Chemotherapy
Drug: MEC (Mitoxantrone, Etoposide, Cytarabine) — IV injection
  Arms: Salvage Chemotherapy
Drug: FLAG-IDA (Granulocyte-Colony Stimulating Factor (G-CSF), Fludarabine, Cytarabine, Idarubicin) — SC (G-CSF) and IV (Fludarabine, Cytarabine, Idarubicin) injection
  Arms: Salvage Chemotherapy

SUMMARY:
The purpose of this study was to determine the clinical benefit of ASP2215 therapy in participants with FMS-like tyrosine kinase (FLT3) mutated acute myeloid leukemia (AML) who were refractory to or had relapsed after first-line AML therapy as shown with overall survival (OS) compared to salvage chemotherapy, and determined the efficacy of ASP2215 therapy as assessed by the rate of complete remission and complete remission with partial hematological recovery (CR/CRh) in these participants. This study also determined the overall efficacy in event-free survival (EFS) and complete remission (CR) rate of ASP2215 compared to salvage chemotherapy.

DETAILED DESCRIPTION:
Participants considered an adult according to local regulations at the time of signing informed consent participated in this study. Participants were randomized in a 2:1 ratio to receive ASP2215 or salvage chemotherapy. Participants entered the screening period up to 14 days prior to the start of treatment. Prior to randomization, a salvage chemotherapy regimen was pre-selected for each participant; options included low-dose cytarabine (LoDAC), azacitidine, mitoxantrone, etoposide, and intermediate-dose cytarabine (MEC), or fludarabine, cytarabine, and granulocyte colony-stimulating factor (G-CSF) with idarubicin (FLAG-IDA). The randomization was stratified by response to first-line therapy and pre-selected salvage chemotherapy. Participants were administered treatment over continuous 28-day cycles. After treatment discontinuation, participants had a pre-hematopoietic stem cell transplant (HSCT)/end-of-treatment visit within 7 days after treatment discontinuation, followed by a 30-day follow-up for safety, in which a telephone contact with the participant was sufficient unless any assessment had to be repeated for resolution of treatment-related adverse events (AEs). After that, long term follow-up was done every 3 months up to 3 years from the participant's end-of-treatment visit.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a diagnosis of primary acute myeloid leukemia (AML) or AML secondary to myelodysplastic syndrome (MDS) according to WHO classification (2008) as determined by pathology review at the treating institute.
* Participant is refractory to or relapsed after first-line AML therapy (with or without hematopoietic stem cell transplant (HSCT)).

  * Refractory to first-line AML therapy is defined as:

    1. Participant did not achieve complete remission/complete remission with incomplete hematologic recovery/complete remission with incomplete platelet recovery (CR/CRi/CRp) under initial therapy. A Participant eligible for standard therapy must receive at least one cycle of an anthracycline containing induction block in standard dose for the selected induction regimen. A Participant not eligible for standard therapy must have received at least one complete block of induction therapy seen as the optimum choice of therapy to induce remission for this subject.
  * Untreated first hematologic relapse is defined as:

    1. Participant must have achieved a CR/CRi/CRp (criteria as defined by [Cheson et al, 2003], see Section 5.3) with first line treatment and has hematologic relapse.
* Participant is positive for FLT3 mutation in bone marrow or whole blood as determined by the central lab. A Participant with rapidly proliferative disease and unable to wait for the central lab results can be enrolled based on a local test performed after completion of the last interventional treatment. Participants can be enrolled from a local test result if they have any of the following FLT3 mutations: FLT3 internal tandem duplication (ITD), FLT3 tyrosine kinase domain (TKD)/D835 or FLT3- TKD/I836.
* Participant has an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* Participant is eligible for pre-selected salvage chemotherapy.
* Participant must meet the following criteria as indicated on the clinical laboratory tests:

  * Serum aspartate aminotransferase and alanine aminotransferase ≤ 2.5 x upper limit of normal (ULN)
  * Serum total bilirubin ≤ 1.5 x ULN
  * Serum creatinine ≤ 1.5 x ULN or an estimated glomerular filtration rate of > 50 mL/min as calculated by the Modification of Diet in Renal Disease equation.
* Participant is suitable for oral administration of study drug.
* Female Participant must either:

  * Be of non-child bearing potential:

    1. post-menopausal (defined as at least 1 year without any menses) prior to Screening, or
    2. documented as surgically sterile (at least 1 month prior to Screening)
  * Or, if of childbearing potential,

    1. Agree not to try to become pregnant during the study and for 180 days after the final study administration
    2. And have a negative urine pregnancy test at Screening
    3. And, if heterosexually active, agree to consistently use highly effective contraception per locally accepted standards in addition to a barrier method starting at Screening and throughout the study period and for 180 days after the final study drug administration.
* Female Participant must agree not to breastfeed at Screening and throughout the study period and for 60 days after the final study drug administration.
* Female Participant must not donate ova starting at Screening and throughout the study period and for 180 days after the final study drug administration.
* Male Participant and their female partners who are of childbearing potential must be using highly effective contraception per locally accepted standards in addition to a barrier method starting at Screening and continue throughout the study period and for 120 days after the final study drug administration.
* Male Participant must not donate sperm starting at Screening and throughout the study period and 120 days after the final study drug administration.
* Participant agrees not to participate in another interventional study while on treatment.

Exclusion Criteria:

* Participant was diagnosed as acute promyelocytic leukemia (APL).
* Participant has BCR-ABL-positive leukemia (chronic myelogenous leukemia in blast crisis).
* Participant has AML secondary to prior chemotherapy for other neoplasms (except for MDS).
* Participant is in second or later hematologic relapse or has received salvage therapy for refractory disease
* Participant has clinically active central nervous system leukemia.
* Participant has been diagnosed with another malignancy, unless disease-free for at least 5 years. Participants with treated nonmelanoma skin cancer, in situ carcinoma or cervical intraepithelial neoplasia, regardless of the disease-free duration, are eligible for this study if definitive treatment for the condition has been completed. Participants with organ-confined prostate cancer with no evidence of recurrent or progressive disease are eligible if hormonal therapy has been initiated or the malignancy has been surgically removed or treated with definitive radiotherapy.
* Participant has received prior treatment with ASP2215 or other FLT3 inhibitors (with the exception of sorafenib and midostaurin used in first-line therapy regimen as part of induction, consolidation, and/or maintenance).
* Participant has clinically significant abnormality of coagulation profile, such as disseminated intravascular coagulation (DIC).
* Participant has had major surgery within 4 weeks prior to the first study dose.
* Participant has radiation therapy within 4 weeks prior to the first study dose.
* Participant has congestive heart failure New York Heart Association (NYHA) class 3 or 4, or Participant with a history of congestive heart failure NYHA class 3 or 4 in the past, unless a screening echocardiogram performed within 3 months prior to study entry results in a left ventricular ejection fraction that is ≥ 45%.
* Participant requires treatment with concomitant drugs that are strong inducers of cytochrome P450 (CYP)3A.
* Participants with mean of triplicate Fridericia-corrected QT interval (QTcF) > 450 ms at Screening based on central reading.
* Participants with Long QT Syndrome at Screening.
* Participants with hypokalemia and hypomagnesemia at Screening (defined as values below lower limit of normal [LLN]).
* Participant requires treatment with concomitant drugs that are strong inhibitors or inducers of P glycoprotein (P-gp) with the exception of drugs that are considered absolutely essential for the care of the subject.
* Participant requires treatment with concomitant drugs that target serotonin 5-hydroxytryptamine receptor 1 (5HT1R) or 5-hydroxytryptamine receptor 2B (5HT2BR) or sigma nonspecific receptor with the exception of drugs that are considered absolutely essential for the care of the subject.
* Participant has an active uncontrolled infection.
* Participant is known to have human immunodeficiency virus infection.
* Participant has active hepatitis B or C, or other active hepatic disorder.
* Participant has any condition which makes the Participant unsuitable for study participation.
* Participant has active clinically significant GVHD or is on treatment with systemic corticosteroids for GVHD.
* Participant has an FLT3 mutation other than the following: FLT3-ITD, FLT3-TKD/D835 or FLT3-TKD/I836.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 371 (Actual)
Dates: Start 2015-10-20 (Actual); Primary Completion 2018-09-17 (Actual); Study Completion 2025-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Executive Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (126):
- United States (37):
  - Site US10011, Birmingham, Alabama
  - Site US10012, Los Angeles, California
  - Site US10076, Orange, California
  - Site US10073, San Francisco, California
  - Site US10067, New Haven, Connecticut
  - Site US10045, Gainesville, Florida
  - Site US10081, Atlanta, Georgia
  - Site US10006, Chicago, Illinois
  - Site US10075, Westwood, Kansas
  - Site US10074, Louisville, Kentucky
  - Site US10048, New Orleans, Louisiana
  - Site US10005, Baltimore, Maryland
  - Site US10034, Boston, Massachusetts
  - Site US10022, Boston, Massachusetts
  - Site US10085, Boston, Massachusetts
  - Site US10087, Detroit, Michigan
  - Site US10057, Minneapolis, Minnesota
  - Site US10023, Lebanon, New Hampshire
  - Site US10027, Hackensack, New Jersey
  - Site US10077, New Brunswick, New Jersey
  - Site US10001, Buffalo, New York
  - Site US10037, New York, New York
  - Site US10008, New York, New York
  - Site US10013, New York, New York
  - Site US10072, New York, New York
  - Site US10046, Syracuse, New York
  - Site US10024, Durham, North Carolina
  - Site US10078, Winston-Salem, North Carolina
  - Site US10044, Cleveland, Ohio
  - Site US10084, Columbus, Ohio
  - Site US10058, Oklahoma City, Oklahoma
  - Site US10041, Hershey, Pennsylvania
  - Site US10010, Philadelphia, Pennsylvania
  - Site US10080, Philadelphia, Pennsylvania
  - Site US10014, Charleston, South Carolina
  - Site US10063, Nashville, Tennessee
  - Site US10035, Milwaukee, Wisconsin
- Site BE32002, Yvoir, Belgium
- Canada (4):
  - Site CA15004, Edmonton, Alberta
  - Site CA15001, Hamilton, Ontario
  - Site CA15015, Toronto, Ontario
  - Site CA15003, Montreal, Quebec
- France (6):
  - Site FR33013, Brest
  - Site FR33002, Le Chesnay
  - Site FR33010, Lille
  - Site FR33009, Pessac
  - Site FR33014, Rennes
  - Site FR33008, Toulouse
- Germany (5):
  - Site DE49009, Dresden
  - Site DE49011, Leipzig
  - Site DE49003, Marburg
  - Site DE49002, München
  - Site DE49010, Tübingen
- Israel (6):
  - Site IL97201, Ashkelon
  - Site IL97209, Haifa
  - Site IL97203, Jerusalem
  - Site IL97210, Jerusalem
  - Site IL97206, Petah Tikva
  - Site IL97208, Rehovot
- Italy (7):
  - Site IT39005, Bologna
  - Site IT39010, Brescia
  - Site IT39001, Milan
  - Site IT39004, Palermo
  - Site IT39011, Pavia
  - Site IT39007, Roma
  - Site IT39002, Varese
- Japan (23):
  - Site JP81002, Nagoya, Aichi-ken
  - Site JP81010, Narita, Chiba
  - Site JP81026, Yoshida-gun, Fukui
  - Site JP81016, Sapporo, Hokkaido
  - Site JP81018, Kobe, Hyōgo
  - Site JP81017, Tsukuba, Ibaraki
  - Site JP81009, Isehara, Kanagawa
  - Site JP81006, Yokohama, Kanagawa
  - Site JP81012, Sendai, Miyagi
  - Site JP81007, Kurashiki, Okayama-ken
  - Site JP81014, Sayama, Osaka
  - Site JP81020, Kawagoe, Saitama
  - Site JP81027, Shimotsuke, Tochigi
  - Site JP81005, Chuo-ku, Tokyo
  - Site JP81004, Shinagawa-ku, Tokyo
  - Site JP81022, Shinjuku-ku, Tokyo
  - Site JP81023, Akita
  - Site JP81021, Aomori
  - Site JP81013, Kumamoto
  - Site JP81025, Kyoto
  - Site JP81008, Nagasaki
  - Site JP81024, Okayama
  - Site JP81011, Osaka
- Poland (3):
  - Site PL48002, Gdansk
  - Site PL48005, Opole
  - Site PL48004, Wroclaw
- South Korea (10):
  - Site KR82005, Suwon, Gyeonggi-do
  - Site KR82010, Busan
  - Site KR82009, Goyang
  - Site KR82003, Jeollanam-do
  - Site KR82007, Seoul
  - Site KR82004, Seoul
  - Site KR82001, Seoul
  - Site KR82002, Seoul
  - Site KR82008, Seoul
  - Site KR82011, Seoul
- Spain (8):
  - Site ES34009, Badalona
  - Site ES34011, Barcelona
  - Site ES34012, Barcelona
  - Site ES34010, Barcelona
  - Site ES34016, Girona
  - Site ES34005, L'Hospitalet de Llobregat
  - Site ES34014, Salamanca
  - Site ES34017, Valencia
- Taiwan (10):
  - Site TW88606, Kaohsiung City
  - Site TW88604, Kaohsiung City
  - Site TW88608, Taichung
  - Site TW88609, Taichung
  - Site TW88601, Tainan
  - Site TW88603, Taipei
  - Site TW88610, Taipei
  - Site TW88611, Taipei
  - Site TW88602, Taipei
  - Site TW88605, Taoyuan District
- Turkey (Türkiye) (2):
  - Site TR90001, Ankara
  - Site TR90004, Ankara
- United Kingdom (4):
  - Site GB44014, Bournemouth
  - Site GB44013, Harrow
  - Site GB44003, Manchester
  - Site GB44015, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Ritchie EK, Cella D, Fabbiano F, Pigneux A, Kanda Y, Ivanescu C, Pandya BJ, Shah MV. Patient-reported outcomes from the phase 3 ADMIRAL trial in patients with FLT3-mutated relapsed/refractory AML. Leuk Lymphoma. 2023 May;64(5):938-950. doi: 10.1080/10428194.2023.2186731. Epub 2023 Apr 5. PMID 37019445
- [Derived] Smith CC, Levis MJ, Perl AE, Hill JE, Rosales M, Bahceci E. Molecular profile of FLT3-mutated relapsed/refractory patients with AML in the phase 3 ADMIRAL study of gilteritinib. Blood Adv. 2022 Apr 12;6(7):2144-2155. doi: 10.1182/bloodadvances.2021006489. PMID 35130342
- [Derived] Perl AE, Larson RA, Podoltsev NA, Strickland S, Wang ES, Atallah E, Schiller GJ, Martinelli G, Neubauer A, Sierra J, Montesinos P, Recher C, Yoon SS, Hosono N, Onozawa M, Chiba S, Kim HJ, Hasabou N, Lu Q, Tiu R, Levis MJ. Follow-up of patients with R/R FLT3-mutation-positive AML treated with gilteritinib in the phase 3 ADMIRAL trial. Blood. 2022 Jun 9;139(23):3366-3375. doi: 10.1182/blood.2021011583. PMID 35081255
- [Derived] Perl AE, Martinelli G, Cortes JE, Neubauer A, Berman E, Paolini S, Montesinos P, Baer MR, Larson RA, Ustun C, Fabbiano F, Erba HP, Di Stasi A, Stuart R, Olin R, Kasner M, Ciceri F, Chou WC, Podoltsev N, Recher C, Yokoyama H, Hosono N, Yoon SS, Lee JH, Pardee T, Fathi AT, Liu C, Hasabou N, Liu X, Bahceci E, Levis MJ. Gilteritinib or Chemotherapy for Relapsed or Refractory FLT3-Mutated AML. N Engl J Med. 2019 Oct 31;381(18):1728-1740. doi: 10.1056/NEJMoa1902688. PMID 31665578
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website — https://www.clinicaltrials.astellas.com/study/2215-CL-0301
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=14515&tenant=MT_AST_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from approximately 140 centers in North America, Europe, Asia and the rest of the world and randomized in a 2:1 ratio to receive gilteritinib or salvage chemotherapy. Participants had FMS-like tyrosine kinase 3 (FLT3) mutations and relapsed or refractory acute myeloid leukemia (AML) after first-line therapy.
Pre-assignment Details: Participants entered the screening period up to 14 days prior to the start of treatment. Prior to randomization, the investigator preselected a salvage chemotherapy for each participant. The randomization was stratified by response to first-line AML therapy and preselected salvage chemotherapy. Treatment was given over continuous 28-day cycles.
Groups:
- Gilteritinib: Participants received 120 mg dose (3 tablets of 40 mg) orally once a day in continuous 28-day cycles, at least 2 hours after or 1 hour before food. Gilteritinib treatment continued until participants met one of the treatment discontinuation criteria. After the end of treatment period, participants were allowed to enter long-term follow up period for up to 3 years for collection of subsequent AML treatment, EuroQol Group-5 Dimension-5 Level Instrument (EQ-5D-5L), remission status and survival (cause of death and date of death). Participants continuing to derive clinical benefit from gilteritinib as assessed by the investigator were allowed to continue the study treatment until a discontinuation criterion was met or if they had completed more than 3 years of treatment.
- Salvage Chemotherapy: Participants received chemotherapy in 28-day cycles. Participants on Low-Dose Cytarabine (LoDAC) received 20 mg of cytarabine twice daily by subcutaneous (SC) or intravenous (IV) injection for 10 days. Participants on azacitidine received 75 mg/m^2 daily by SC or IV injection for 7 days. Participants on LoDAC or azacitidine treatment continued until they met discontinuation criteria. Participants on mitoxantrone, etoposide and intermediate-dose cytarabine (MEC) chemotherapy received mitoxantrone 8 mg/m^2 daily by IV for 5 days, etoposide 100 mg/m^2 daily by IV for 5 days and cytarabine 1000 mg/m^2 daily by IV for 5 days (days 1-5). Participants on fludarabine, cytarabine and granulocyte colony-stimulating factor with idarubicin (FLAG-IDA) chemotherapy received granulocyte-colony stimulating factor (G-CSF) 300 μg/m^2 daily by SC/IV for 5 days (days 1-5), fludarabine 30 mg/m^2 daily by IV for 5 days (days 2-6), cytarabine 2000 mg/m^2 daily by IV for 5 days (days 2-6) and idarubicin 10 mg/m^2 daily by IV for 3 days (days 2-4). Participants receiving MEC or FLAG-IDA received 1 cycle of therapy and were assessed for response on or after day 15. After the end of treatment period, participants were allowed to enter the long-term follow-up period of up to 3 years for collection of subsequent AML treatment, EQ-5D-5L, remission status and survival (cause of death and date of death).
Period: Randomization Period: Up to 3 Years
Arm/Group | Gilteritinib | Salvage Chemotherapy
Started | 247 | 124
Treated | 246 | 109
Completed | 0 | 19
Not Completed | 247 | 105
Not completed — Progressive disease | 76 | 16
Not completed — Lack of Efficacy | 21 | 31
Not completed — Death | 38 | 10
Not completed — Disease relapse | 37 | 2
Not completed — Adverse Event | 32 | 5
Not completed — Withdrawal by Subject | 9 | 24
Not completed — Physician Decision | 13 | 11
Not completed — Protocol deviation | 1 | 1
Not completed — Miscellaneous | 20 | 5
Period: Long Term Follow up: up to 3 Years
Arm/Group | Gilteritinib | Salvage Chemotherapy
Started | 133 | 73
Completed | 0 | 0
Not Completed | 133 | 73
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Lost to Follow-up | 1 | 2
Not completed — Death | 118 | 65
Not completed — Miscellaneous | 10 | 1

BASELINE CHARACTERISTICS:
Population: The analysis population was the Intention to Treatment (ITT), which consisted of all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Gilteritinib | Salvage Chemotherapy | Total
Number analyzed (Participants) | 247 | 124 | 371
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59 (14.6) | 57.6 (14.8) | 58.5 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 131 | 70 | 201
  Male | 116 | 54 | 170
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  WHITE | 145 | 75 | 220
  ASIAN | 69 | 33 | 102
  BLACK OR AFRICAN AMERICAN | 14 | 7 | 21
  NATIVE HAWAIIAN OR OTHER PACIFIC ISLANDER | 1 | 0 | 1
  AMERICAN INDIAN OR ALASKA NATIVE | 0 | 0 | 0
  UNKNOWN | 4 | 4 | 8
  OTHER | 5 | 1 | 6
  MISSING | 9 | 4 | 13
Ethnicity [Count of Participants; unit: Participants]
  NOT HISPANIC OR LATINO | 221 | 116 | 337
  HISPANIC OR LATINO | 12 | 2 | 14
  UNKNOWN | 3 | 2 | 5
  MISSING | 11 | 4 | 15
Cytogenic Risk Status [Count of Participants; unit: Participants] — The category of "Other" includes those with cytogenetic risk status that cannot be categorized as favorable, intermediate or unfavorable.
  Participants
    INTERMEDIATE | 182 | 89 | 271
    UNFAVORABLE | 26 | 11 | 37
    FAVORABLE | 4 | 1 | 5
    OTHER | 35 | 23 | 58
Baseline Eastern Cooperative Oncology Group (ECOG) [Count of Participants; unit: Participants] — ECOG performance status is a scale used to assess impact on daily activities. It is based on the investigator assessment. Scores range from 0 to 5, with 0-signifying fully active participant; 1-restricted in physically strenuous activity; 2-ambulatory and capable of all self-care, unable to work; 3-capable of only limited self-care, confined to bed more than 50% of waking hours; 4-completely disabled and 5-dead. Negative numerical score indicates an improvement and positive numerical score indicates a decline in participant's daily activities, indicating disease progression.
  Participants
    0-1 | 206 | 105 | 311
    >=2 | 41 | 19 | 60
FLT3 Mutation Status by Central Testing by FLT3 CDx [Count of Participants; unit: Participants]
  FLT3-ITD Alone | 215 | 113 | 328
  FLT3-TKD Alone | 21 | 10 | 31
  FLT3-ITD and FLT3-TKD | 7 | 0 | 7
  Others (Unknown/Missing/Negative) | 4 | 1 | 5
Prior Use of FLT3 Inhibitor [Count of Participants; unit: Participants] — Prior use of FLT3 inhibitor is defined as 'Yes' if participants received prior AML therapy of midostaurin, sorafenib or quizartinib; otherwise, prior use of FLT3 inhibitor is assigned as No.
  Participants
    No | 215 | 110 | 325
    Yes | 32 | 14 | 46
Region [Count of Participants; unit: Participants]
  NORTH AMERICA | 114 | 52 | 166
  EUROPE | 68 | 43 | 111
  ASIA | 65 | 29 | 94
Baseline Body Surface Area (BSA) [Mean (Standard Deviation); unit: m^2] — Population: The analysis population was the ITT, with available data.
  m^2
    number analyzed (Participants) | 199 | 122 | 321
    (all) | 1.815 (0.281) | 1.777 (0.257) | 1.8 (0.272)
Baseline Height [Mean (Standard Deviation); unit: centimeter (cm)] — Population: The analysis population was the ITT, with available data.
  centimeter (cm)
    number analyzed (Participants) | 234 | 123 | 357
    (all) | 167.25 (10.31) | 166.39 (10.63) | 166.95 (10.41)
Baseline Weight [Mean (Standard Deviation); unit: kilogram (kg)] — Population: The analysis population was the ITT, with available data.
  kilogram (kg)
    number analyzed (Participants) | 243 | 124 | 367
    (all) | 72.79 (20.47) | 69.91 (19.73) | 71.82 (20.25)
Response to First Line Therapy [Count of Participants; unit: Participants] — Baseline stratification factors.
  Participants
    Primary refractory without HSCT | 98 | 48 | 146
    Relapse within 6 months after CRc and no HSCT | 67 | 34 | 101
    Relapse after 6 months after CRc and no HSCT | 34 | 17 | 51
    Relapse within 6 months after allogeneic HSCT | 31 | 17 | 48
    Relapse after 6 months after allogeneic HSCT | 17 | 8 | 25
Preselected Salvage Chemotherapy [Count of Participants; unit: Participants] — Baseline stratification factors.
  Participants
    High intensity chemotherapy | 149 | 75 | 224
    Low intensity chemotherapy | 98 | 49 | 147
Response to First Line Therapy-Preselected Salvage Chemotherapy [Count of Participants; unit: Participants] — Baseline stratification factors. HSCT is hematopoietic stem cell transplant. CRc is composite complete remission.
  Participants
    Primary refractory w/o HSCT, high intensity (IT) | 57 | 28 | 85
    Primary refractory w/o HSCT, low IT | 41 | 20 | 61
    Relapse w/I 6 mths after CRc and no HSCT, high IT | 40 | 21 | 61
    Relapse w/I 6 mths after CRc and no HSCT low IT | 27 | 13 | 40
    Relapse after 6 mths after CRc and no HSCT high IT | 23 | 11 | 34
    Relapse w/I 6 mths after allogeneic HSCT low IT | 16 | 9 | 25
    Relapse w/I 6 mths after allogeneic HSCT high IT | 15 | 8 | 23
    Relapse after 6 mths after allogeneic HSCT high IT | 14 | 7 | 21
    Relapse after 6 mths after CRc and no HSCT low IT | 11 | 6 | 17
    Relapse after 6 mths after allogeneic HSCT low IT | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Duration of Overall Survival (OS)
Description: Overall survival was defined as the time from the date of randomization until the date of death from any cause (death date - randomization date + 1). For a participant who was not known to have died by the end of study follow-up, OS was censored at the date of last contact (date of last contact - randomized date + 1). The date of last contact was the latest date that the participant was known to be alive. The last contact date was derived for participants alive at the analysis cutoff date. Survival rate and 95% CI were estimated using the Kaplan-Meier method and the Greenwood formula.
Time Frame: From randomization to until the date of death from any cause (median time of follow-up for OS was 17.8 months)
Population: The analysis population was the Intention to Treatment (ITT) which consisted of all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Gilteritinib | Salvage Chemotherapy
Number analyzed (Participants) | 247 | 124
Months | 9.3 [7.7 to 10.7] | 5.6 [4.7 to 7.3]
Statistical Analysis 1: Comparison: Gilteritinib vs Salvage Chemotherapy; Stratified analysis where tratification factors were response to first-line AML therapy and preselected salvage chemotherapy per IRT; Test type: Other; p = 0.0004, Log Rank — 1-sided P-value; Hazard Ratio (HR) = 0.637, 95% CI 2-sided [0.490 to 0.830] — Based on Cox proportional hazards model. Assuming proportional hazards, an HR of < 1 indicates a reduction in the hazard rate in favor of the gilteritinib arm

2. Primary Outcome: Percentage of Participants With Complete Remission and Complete Remission With Partial Hematological Recovery (CR/CRh) in the Gilteritinib Arm
Description: The CR/CRh rate was defined as the number of participants who achieved either CR or CRh divided by the number of participants in the analysis population.
  CR: For participants to be classified as being in CR at, they must have had bone marrow regenerating normal hematopoietic cells and achieved a morphologic leukemia-free state and must had an ANC ≥ 1 x 10^9/L and platelet count ≥ 100 x 10^9/L and normal marrow differential with < 5% blasts, and they were RBC and platelet transfusion independent (defined as 1 week without RBC transfusion and 1 week without platelet transfusion). There was no evidence of extramedullary leukemia.
  CRh: Participants were classified as CRh if they had marrow blasts < 5%, partial hematologic recovery ANC ≥ 0.5 x 10^9/L and platelets ≥ 50 x 10^9/L, no evidence of extramedullary leukemia and could not be classified as CR.
Time Frame: From the date of randomization up to at least 112 days
Population: The analysis population was the response analysis set (RAS) which consisted of participants who were who were at least 112 days past the first dose of gilteritinib or randomization (for participants who did not receive gilteritinib). The participants were analyzed based on the randomized treatments.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Gilteritinib
Number analyzed (Participants) | 142
Percentage of participants
  CR/CRh rate | 28.2 [20.9 to 36.3]
  CR rate | 19.0 [12.9 to 26.4]
  CRh rate | 9.2 [5.0 to 15.1]

3. Secondary Outcome: Duration of Event-Free Survival (EFS)
Description: EFS: time from randomization date up to date of documented relapse (excluding relapse after PR)/ treatment failure (failure to achieve CR, CRp, CRi /PR) /death, whichever occurred first. Relapse: leukemic blasts in peripheral blood 5/ ≥ 25% blasts in bone marrow (BM) aspirate due to no other cause/reappearance/new appearance of extramedullary leukemia. CR: BM regenerating normal hematopoietic cells, morphologic leukemia-free state, ANC ≥1x10^9/L, platelet count ≥100x10^9/L, normal marrow differential with <5% blasts, and RBC/platelet transfusion independent with no extramedullary leukemia. CRp: achieved CR except incomplete platelet recovery (<100x 0^9/L). CRi: criteria for CR fulfilled except incomplete hematological recovery with residual neutropenia <1x10^9/L with /without complete platelet recovery. PR: BM regenerating normal hematopoietic cells, peripheral recovery, no circulating blasts and decrease of 50% blasts in with total blasts between 5% -25% or, 5% if Auer rods present.
Time Frame: From the date of randomization until the date of documented relapse, treatment failure or death from any cause (median time of follow-up was 17.8 months)
Population: The analysis population was the ITT with available data.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Gilteritinib | Salvage Chemotherapy
Number analyzed (Participants) | 189 | 62
Months | 2.8 [1.4 to 3.7] | 0.7 [0.2 to NA] — Not estimable. Data could not be estimated due to low number of events.
Statistical Analysis 1: Comparison: Gilteritinib vs Salvage Chemotherapy; Stratification factors were response to first-line AML therapy and preselected salvage chemotherapy per IRT; Test type: Other; p = 0.0415, Log Rank — 1-sided P-value; Hazard Ratio (HR) = 0.793, 95% CI 2-sided [0.577 to 1.089] — Based on the Cox proportional hazards model. Assuming proportional hazards, an HR of < 1 indicates a reduction in the hazard rate in favor of the gilteritinib arm

4. Secondary Outcome: Percentage of Participants With Complete Remission (CR) Rate
Description: The CR rate was defined as the number of participants who achieved the best response of CR divided by the number of participants in the analysis population. CR: For participants to be classified as being in CR, they must have had bone marrow regenerating normal hematopoietic cells and achieved a morphologic leukemia-free state and must had an ANC ≥ 1 x 10^9/L and platelet count ≥ 100 x 10^9/L and normal marrow differential with < 5% blasts, and they were RBC and platelet transfusion independent (defined as 1 week without RBC transfusion and 1 week without platelet transfusion). There was no evidence of extramedullary leukemia.
Time Frame: From the date of randomization up to at least 6 months
Population: The analysis population was the ITT.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Gilteritinib | Salvage Chemotherapy
Number analyzed (Participants) | 247 | 124
Percentage of participants | 21.1 [16.1 to 26.7] | 10.5 [5.7 to 17.3]
Statistical Analysis 1: Comparison: Gilteritinib vs Salvage Chemotherapy; Based on stratified Cochran-Mantel-Haenszel test. Stratification factors were response to first-line AML therapy and preselected salvage chemotherapy per IRT. Treatment difference = gilteritinib -chemotherapy; Test type: Other; p = 0.0106, Cochran-Mantel-Haenszel — Stratified P-value; Adjusted Treatment Difference = 10.6, 95% CI 2-sided [2.8 to 18.4]

5. Secondary Outcome: Duration of Leukemia-Free Survival (LFS)
Description: LFS: time from the date of first CRc until the date of documented relapse or death for subjects who achieve CRc. For a subject who is not known to have relapsed or died, LFS is censored on the date of last relapse-free disease assessment date. CRc: achieved CR, CRp or CRi. Relapse: leukemic blasts in peripheral blood/ ≥ 25% blasts in bone marrow (BM) aspirate not due to any other cause/reappearance/new appearance of extramedullary leukemia. CR: BM regenerating normal hematopoietic cells, morphologic leukemia-free state, ANC ≥ 1 x 10^9/L, platelet count ≥ 100 x 10^9/L, normal marrow differential with < 5% blasts, and RBC/platelet transfusion independent with no extramedullary leukemia. CRp: achieved CR except incomplete platelet recovery (< 100 x 10^9/L). CRi : criteria for CR fulfilled except incomplete hematological recovery with residual neutropenia < 1 x 10^9/L with /without complete platelet recovery..
Time Frame: From the date of first CRc until the date of documented relapse or death for participants who achieved CRc (median time of follow-up was 17.8 months)
Population: The analysis population was the ITT, with participants with best response of CRc.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Gilteritinib | Salvage Chemotherapy
Number analyzed (Participants) | 134 | 27
Months | 4.4 [3.6 to 5.2] | 6.7 [2.1 to 8.5]
Statistical Analysis 1: Comparison: Gilteritinib vs Salvage Chemotherapy; The LFS was analyzed for participants who achieved remission using the stratified log-rank test with strata to control for response to first-line AML therapy and preselected salvage chemotherapy. Duration of LFS was based on Kaplan-Meier estimates; Test type: Other; p = 0.6654, Log Rank — Unstratified p-value; Hazard Ratio (HR) = 0.889, 95% CI 2-sided [0.506 to 1.563] — [estimate comment as in outcome 3, analysis 1]

6. Secondary Outcome: Duration of Remission
Description: Duration of remission included duration of CRc, CR/CRh, CRh, CR, CRi, CRp (defined as the time from the date of first CRc until the date of first documented relapse for participants who achieved CRc, CR/CRh, CRh, CR, CRi, CRp respectively) and duration of response (CRc + PR). CRc: achieved CR, CRp or CRi at the visit. CR: BM regenerating normal hematopoietic cells, morphologic leukemia-free state, ANC ≥1x10^9/L, platelet count ≥100x10^9/L, normal marrow differential with <5% blasts, and RBC/platelet transfusion independent with no extramedullary leukemia. CRp: achieved CR except incomplete platelet recovery (<100x 0^9/L). CRi: criteria for CR fulfilled except incomplete hematological recovery with residual neutropenia <1x10^9/L with /without complete platelet recovery. PR: BM regenerating normal hematopoietic cells, peripheral recovery, no circulating blasts and decrease of 50% blasts in with total blasts between 5% -25% or, 5% if Auer rods present.
Time Frame: From the date of first response until the date of documented relapse for participants who achieved CRc or PR (median time of follow-up was 17.8 months)
Population: The analysis population was the ITT, Duration of CR was only applicable to participants with best overall response of CR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Gilteritinib | Salvage Chemotherapy
Number analyzed (Participants) | 52 | 13
Months | 14.8 [11.0 to NA] — Not estimable. Data could not be estimated due to low number of events. | 1.8 [NA to NA] — Not estimable. Data could not be estimated due to low number of events.
Statistical Analysis 1: Comparison: Gilteritinib vs Salvage Chemotherapy; Test type: Other; p = 0.1189, Log Rank — Unstratified; Hazard Ratio (HR) = 0.206, 95% CI 2-sided [0.022 to 1.886] — Based on Cox proportional hazards model. Assuming proportional hazards, a hazard ratio < 1 indicates a reduction in hazard rate in favor of gilteritinib arm

7. Secondary Outcome: Percentage of Participants With Composite Complete Remission (CRc Rate)
Description: CRc rate: Number of participants with best response of CRc (CR,complete remission with incomplete platelet recovery [CRp] or complete remission with incomplete hematologic recovery [CRi]) divided by number of participants in the analysis population. CRc : Participants who achieved CR, CRp or CRi at a post-baseline visit. CR: Participants having bone marrow regenerating normal hematopoietic cells, a morphologic leukemia-free state, an ANC ≥ 1 x 10^9/L and platelet count ≥ 100 x 10^9/L, normal marrow differential with < 5% blasts, and being RBC and platelet transfusion independent with no evidence of extramedullary leukemia at a post-baseline visit. CRp: Participants achieving CR except for incomplete platelet recovery (< 100 x 10^9/L) at a post-baseline visit. CRi : Participants, who fulfilled all criteria for CR except incomplete hematological recovery with residual neutropenia < 1 x 10^9/L with or without complete platelet recovery at a post-baseline visit.
Time Frame: From the date of randomization up to at least 6 months
Population: The analysis population was the ITT.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Gilteritinib | Salvage Chemotherapy
Number analyzed (Participants) | 247 | 124
Percentage of participants | 54.3 [47.8 to 60.6] | 21.8 [14.9 to 30.1]
Statistical Analysis 1: Comparison: Gilteritinib vs Salvage Chemotherapy; Treatment difference = gilteritinib - chemotherapy. The 95% CIs were asymptotic confidence limits using the normal approximation to the binomial distribution; Test type: Other; p < 0.0001, 2-sided Fisher's exact test — Unstratified 2-sided P-value; Treatment difference = 32.5, 95% CI 2-sided [22.3 to 42.6]

8. Secondary Outcome: Percentage of Participants Who Underwent Hematopoietic Stem Cell Transplant
Description: Transplantation rate is defined as the percentage of participants undergoing Hematopoietic stem cell transplant (HSCT) during the study period.
Time Frame: From the date of randomization until end of study (median time of follow-up was 17.8 months)
Population: The analysis population is the ITT.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Gilteritinib | Salvage Chemotherapy
Number analyzed (Participants) | 247 | 124
Percentage of participants | 25.5 [20.2 to 31.4] | 15.3 [9.5 to 22.9]
Statistical Analysis 1: Comparison: Gilteritinib vs Salvage Chemotherapy; Test type: Other; p = 0.0333, 2-sided Fisher's exact test — Unstratified 2-sided P-value; Treatment difference = gilteritinib - chemotherapy; Treatment Difference = 10.2, 95% CI 2-sided [1.2 to 19.1]

9. Secondary Outcome: Change From Baseline in Brief Fatigue Inventory (BFI)
Description: The Brief Fatigue Inventory (BFI) was a screening tool designed to assess the severity and impact of fatigue on daily functioning of participants with cancer during the 24 hours. There are 9 items on the scale. The first three questions asked participants to rate their fatigues on a scale from 0 (no fatigue) - 10 (as bad as you can imagine), with higher scores indicating worse outcome. The remaining six questions asked participants to rate how much fatigue has interfered with their daily activities on a scale from 0 (Does not interfere) to 10 (Completely interferes). A global fatigue score can be obtained by averaging all the items on the BFI. The total score range is 0-10 with a higher BFI fatigue score indicates worse outcome. The global BFI score was calculated only if at least 5 of the 9 items are answered.
Time Frame: Baseline, Cycle 1 Day 8 and Cycle 2 Day 1
Population: The analysis population was the ITT, with participants with data at baseline.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Gilteritinib | Salvage Chemotherapy
Number analyzed (Participants) | 227 | 97
Units on a scale
  Cycle 1 day 8 (C1D8): number analyzed (Participants) | 191 | 73
  Cycle 1 day 8 (C1D8) | -0.4 (2.1) | 1.0 (2.3)
  Cycle 2 day 1 (C2D1): number analyzed (Participants) | 206 | 15
  Cycle 2 day 1 (C2D1) | 0.0 (2.6) | 0.4 (2.8)
Statistical Analysis 1: Comparison: Gilteritinib vs Salvage Chemotherapy; C1D8: Using analysis of covariance (ANCOVA) including treatment as a fixed factor, baseline score, response to first-line AML therapy and preselected salvage chemotherapy per IRT as covariates. Least Square (LS) Mean difference was estimated using chemotherapy as control; Test type: Other; p = 0.0000, ANCOVA; Least Squares Mean Difference = -1.2567
Statistical Analysis 2: Comparison: Gilteritinib vs Salvage Chemotherapy; C2D1: Using analysis of covariance (ANCOVA) including treatment as a fixed factor, baseline score, response to first-line AML therapy and preselected salvage chemotherapy per IRT as covariates. Least Square (LS) Mean difference was estimated using chemotherapy as control; Test type: Other; p = 0.8037, ANCOVA; Least Squares Mean Difference = 0.1574

10. Secondary Outcome: Percentage of Participants With Complete Remission (CR) With Partial Hematological Recovery (CRh)
Description: CRh rate was defined as the number of participants who achieved CRh at any of the postbaseline visits and did not have a best response of CR divided by the number of participants in the analysis population.
  CR: For participants to be classified as being in CR at a post-baseline visit, they must have had bone marrow regenerating normal hematopoietic cells and achieved a morphologic leukemia-free state and must had an ANC ≥ 1 x 10^9/L and platelet count ≥ 100 x 10^9/L and normal marrow differential with < 5% blasts, and they were RBC and platelet transfusion independent (defined as 1 week without RBC transfusion and 1 week without platelet transfusion). There was no evidence of extramedullary leukemia.
  CRh: At a post baseline visit, participantss were classified as CRh if they had marrow blasts < 5%, partial hematologic recovery ANC ≥ 0.5 x 10^9/L and platelets ≥ 50 x 10^9/L, no evidence of extramedullary leukemia and could not be classified as CR.
Time Frame: From the date of randomization up to at least 6 months
Population: The analysis population was the ITT.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Gilteritinib | Salvage Chemotherapy
Number analyzed (Participants) | 247 | 124
Percentage of participants | 34.0 [28.1 to 40.3] | 15.3 [9.5 to 22.9]
Statistical Analysis 1: Comparison: Gilteritinib vs Salvage Chemotherapy; Based on a stratified Cochran-Mantel-Haenszel test. Stratification factors were response to first-line AML therapy and preselected salvage chemotherapy per IRT. Pooled strata were used as shown in Table 12.3.3.2. Treatment differences were adjusted based on pooled strata. Treatment difference = gilteritinib 120 mg - chemotherapy; Test type: Other; p < 0.0171, Cochran-Mantel-Haenszel — Stratified 1-sided P-value; Adjusted Treatment Difference, = 18.6, 95% CI 2-sided [9.8 to 27.4]

11. Secondary Outcome: Percentage of Participants Who Achieved Transfusion Conversion and Maintenance
Description: Transfusion conversion & maintenance rate was defined for gilteritinib arm. Participants were classified as transfusion independent if there were no RBC or platelet transfusions within 28 days prior to the first dose to 28 days after the first dose; otherwise they were classified as transfusion dependent at baseline. Participants were considered independent postbaseline if they had 1 consecutive 8 week period without any RBC or platelet transfusion from 29 days after the first dose until the last dose date. For participants who were on treatment ≤ 4 weeks or > 4 weeks but < 12 weeks and there was no RBC or platelet transfusion within postbaseline period, they were considered not evaluable; otherwise, they were considered postbaseline transfusion dependent. Transfusion conversion rate was defined for participants who had evaluable postbaseline transfusion status. Transfusion status (independent vs. dependent) at baseline and postbaseline was reported in a 2 by 2 contingency table.
Time Frame: From 29 days post first dose of study drug until last dose(median treatment duration was (126.00 [4.0, 885.0])
Population: The analysis population was the ITT, with participants who had evaluable postbaseline transfusion status.
Measure: Number; unit: Percentage of participants
Arm/Group | Gilteritinib
Number analyzed (Participants) | 246
Percentage of participants
  Baseline Independent/ Post baseline Independent | 59.2
  Baseline Independent/Post baseline Dependent | 24.5
  Baseline Independent/Post baseline Not Evaluable | 16.3
  Baseline Dependent/Post baseline Independent | 34.5
  Baseline Dependent/Post baseline Dependent | 55.8
  Baseline Dependent/Post baseline Not Evaluable | 9.6

12. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: An AE was defined as any untoward medical occurrence in a participant, temporally associated with the use of study drug, whether or not related to it. It could be any unfavorable/unintended sign (including abnormal laboratory finding), symptom, or disease (new/exacerbated) temporally associated with use of the study drug. A treatment-emergent adverse event (TEAE) : AEs observed after starting administration of study drug (gilteritinib or salvage chemotherapy). Serious AEs (SAEs): AEs which caused death, were life-threatening, resulted in persistent/significant disability/incapacity or disruption of the ability to conduct normal life functions, congenital anomaly, birth defect, required inpatient hospitalization/led to prolongation of hospitalization. Based on national cancer institute common terminology criteria (NCI-CTCAE), AEs were graded as grade 1=mild, grade 2=moderate, grade 3 =severe or medically significant, grade 4 =life threatening, grade 5 =death related to AE
Time Frame: From first dose of study drug up to 30 days after the last dose of study drug (median treatment duration for gilteritinib was (126.00 [4.0, 885.0]) days versus salvage chemotherapy 28.0 [5.0, 217.0] days)
Population: The analysis population was the safety analysis set (SAF), which consisted of participants who received who received at least 1 dose of study drug (gilteritinib or salvage chemotherapy).
Measure: Count of Participants; unit: Participants
Arm/Group | Gilteritinib | Salvage Chemotherapy
Number analyzed (Participants) | 246 | 109
Participants
  Drug-related TEAE | 208 | 71
  Serious TEAE | 211 | 34
  Drug-related serious TEAE | 92 | 16
  TEAE leading to death | 76 | 16
  Drug-related TEAE leading to death | 11 | 5
  TEAE leading to withdrawal of treatment | 65 | 13
  Drug-related TEAE lead withdrawal of treatment | 30 | 5
  NCI-CTCAE Grade 3 or higher TEAE | 238 | 94
  Drug-related Grade 3 or higher TEAE | 157 | 57
  Death | 203 | 87

ADVERSE EVENTS:
Time Frame: Adverse events: From first dose of study drug up to 30 days after the last dose of study drug (median treatment duration for gilteritinib was (126.00 [4.0, 885.0]) days versus salvage chemotherapy 28.0 [5.0, 217.0] days) All cause mortality: From randomization up to end of study (approximately 112 months)
Description: Adverse events: The SAF consisted of all participants who received at least dose of study treatment (gilteritinib or salvage chemotherapy).
  All cause mortality: All randomised participants.
Arm/Group | Gilteritinib | Salvage Chemotherapy
All-Cause Mortality (participants affected / at risk) | 204/247 | 96/124
Serious Adverse Events (participants affected / at risk) | 211/246 | 34/109
Other Adverse Events (participants affected / at risk) | 242/246 | 103/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gilteritinib (N=246) | Salvage Chemotherapy (N=109)
Anaemia (Blood and lymphatic system disorders) | 8 (11) | 0 (0)
Aplasia pure red cell (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 (3) | 0 (0)
Bone marrow failure (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 76 (113) | 9 (15)
Haemolytic anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 3 (4) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac arrest (Cardiac disorders) | 4 (5) | 0 (0)
Cardiac failure (Cardiac disorders) | 3 (3) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 2 (3) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 2 (2) | 0 (0)
Pericardial effusion (Cardiac disorders) | 3 (5) | 0 (0)
Pericardial haemorrhage (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 3 (3) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Accessory breast (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Hamartoma (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Deafness bilateral (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 1 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 11 (14) | 0 (0)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal perforation (Gastrointestinal disorders) | 1 (2) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (2) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 2 (4) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 3 (4) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Stomatitis necrotising (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tongue haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 3 (3) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Face oedema (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 4 (4) | 1 (1)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Mucosal haemorrhage (General disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 2 (2) | 1 (1)
Oedema (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 34 (45) | 1 (2)
Swelling face (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (7) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0)
Acute graft versus host disease in intestine (Immune system disorders) | 1 (2) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 3 (3) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (2) | 0 (0)
Graft versus host disease (Immune system disorders) | 1 (1) | 0 (0)
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 1 (1) | 0 (0)
Abscess bacterial (Infections and infestations) | 1 (1) | 0 (0)
Adenoviral upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 10 (11) | 1 (1)
Bacterial colitis (Infections and infestations) | 1 (2) | 0 (0)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 2 (3) | 0 (0)
Bronchitis (Infections and infestations) | 5 (6) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 2 (4) | 0 (0)
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 6 (6) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 2 (2) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 4 (4) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 1 (2) | 0 (0)
Device related infection (Infections and infestations) | 4 (4) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 1 (2) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 4 (5) | 0 (0)
Epstein-Barr viraemia (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 2 (4) | 0 (0)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 3 (3) | 1 (1)
Eye infection (Infections and infestations) | 1 (1) | 0 (0)
Eye infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Eye infection toxoplasmal (Infections and infestations) | 1 (1) | 0 (0)
Haemophilus infection (Infections and infestations) | 0 (0) | 1 (1)
Hepatic infection (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (3) | 1 (2)
Influenza (Infections and infestations) | 3 (3) | 1 (2)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Large intestine infection (Infections and infestations) | 1 (1) | 0 (0)
Leptotrichia infection (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 2 (3) | 0 (0)
Lower respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection fungal (Infections and infestations) | 2 (2) | 0 (0)
Oesophageal infection (Infections and infestations) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Parotitis (Infections and infestations) | 1 (1) | 0 (0)
Periorbital infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 43 (66) | 8 (12)
Pneumonia fungal (Infections and infestations) | 3 (3) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 2 (2) | 0 (0)
Pseudomonal bacteraemia (Infections and infestations) | 2 (2) | 0 (0)
Pseudomonal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 3 (4) | 0 (0)
Respiratory tract infection (Infections and infestations) | 4 (6) | 0 (0)
Respiratory tract infection fungal (Infections and infestations) | 1 (2) | 0 (0)
Scrotal infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 19 (24) | 7 (11)
Septic shock (Infections and infestations) | 10 (17) | 1 (1)
Sinusitis (Infections and infestations) | 3 (4) | 0 (0)
Sinusitis fungal (Infections and infestations) | 1 (2) | 0 (0)
Skin infection (Infections and infestations) | 4 (7) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 6 (6) | 0 (0)
Staphylococcal infection (Infections and infestations) | 2 (2) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 3 (4) | 0 (0)
Systemic bacterial infection (Infections and infestations) | 2 (3) | 0 (0)
Systemic mycosis (Infections and infestations) | 1 (2) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 5 (6) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection enterococcal (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 2 (3) | 0 (0)
Vulval cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anaphylactic transfusion reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 8 (8) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 13 (17) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 10 (14) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Blood fibrinogen decreased (Investigations) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0)
Blood pressure decreased (Investigations) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 2 (3) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
General physical condition abnormal (Investigations) | 1 (1) | 0 (0)
Liver function test increased (Investigations) | 1 (1) | 0 (0)
Menstruation normal (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 4 (6) | 0 (0)
Norovirus test positive (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 5 (11) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 0 (0)
Adult failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (2) | 1 (2)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hyponatraemic syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 35 (40) | 4 (6)
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (9) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Central nervous system leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Leukaemia cutis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (2)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Soft tissue sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (2)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 2 (2) | 0 (0)
Cerebellar haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 3 (3) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 5 (5) | 0 (0)
Hemiplegia (Nervous system disorders) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 7 (8) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0)
Mania (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 18 (23) | 4 (5)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (2)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Obliterative bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 3 (5)
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 3 (3) | 1 (1)
Haematoma (Vascular disorders) | 4 (6) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 6 (6) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gilteritinib (N=246) | Salvage Chemotherapy (N=109)
Anaemia (Blood and lymphatic system disorders) | 112 (493) | 38 (80)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 8 (9) | 6 (6)
Febrile neutropenia (Blood and lymphatic system disorders) | 57 (73) | 32 (37)
Neutropenia (Blood and lymphatic system disorders) | 32 (115) | 16 (18)
Thrombocytopenia (Blood and lymphatic system disorders) | 62 (301) | 17 (41)
Atrial fibrillation (Cardiac disorders) | 13 (15) | 1 (3)
Tachycardia (Cardiac disorders) | 13 (14) | 7 (7)
Dry eye (Eye disorders) | 27 (28) | 3 (3)
Retinal haemorrhage (Eye disorders) | 20 (23) | 2 (2)
Vision blurred (Eye disorders) | 20 (22) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 37 (44) | 16 (17)
Abdominal pain upper (Gastrointestinal disorders) | 13 (18) | 3 (5)
Constipation (Gastrointestinal disorders) | 77 (96) | 16 (18)
Diarrhoea (Gastrointestinal disorders) | 82 (136) | 32 (37)
Dry mouth (Gastrointestinal disorders) | 22 (23) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 13 (16) | 7 (7)
Mouth ulceration (Gastrointestinal disorders) | 13 (14) | 2 (2)
Nausea (Gastrointestinal disorders) | 83 (129) | 36 (41)
Stomatitis (Gastrointestinal disorders) | 35 (46) | 15 (19)
Vomiting (Gastrointestinal disorders) | 57 (89) | 15 (16)
Asthenia (General disorders) | 35 (49) | 10 (11)
Chills (General disorders) | 23 (33) | 8 (9)
Fatigue (General disorders) | 71 (102) | 14 (17)
Mucosal inflammation (General disorders) | 13 (13) | 9 (11)
Oedema (General disorders) | 15 (18) | 3 (3)
Oedema peripheral (General disorders) | 61 (80) | 13 (19)
Pain (General disorders) | 17 (21) | 1 (1)
Pyrexia (General disorders) | 93 (147) | 31 (57)
Graft versus host disease (Immune system disorders) | 16 (22) | 1 (1)
Cellulitis (Infections and infestations) | 15 (17) | 1 (2)
Nasopharyngitis (Infections and infestations) | 13 (25) | 2 (2)
Oral candidiasis (Infections and infestations) | 13 (14) | 3 (3)
Pneumonia (Infections and infestations) | 40 (46) | 5 (5)
Sinusitis (Infections and infestations) | 15 (21) | 2 (3)
Upper respiratory tract infection (Infections and infestations) | 21 (48) | 3 (3)
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 10 (17) | 7 (13)
Contusion (Injury, poisoning and procedural complications) | 14 (18) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 19 (28) | 1 (1)
Alanine aminotransferase increased (Investigations) | 100 (249) | 10 (20)
Aspartate aminotransferase increased (Investigations) | 97 (253) | 13 (21)
Blood alkaline phosphatase increased (Investigations) | 55 (113) | 2 (2)
Blood bilirubin increased (Investigations) | 21 (68) | 7 (9)
Blood creatine phosphokinase increased (Investigations) | 35 (111) | 0 (0)
Blood creatinine increased (Investigations) | 32 (78) | 4 (4)
Blood lactate dehydrogenase increased (Investigations) | 24 (35) | 5 (5)
Electrocardiogram QT prolonged (Investigations) | 16 (19) | 0 (0)
International normalised ratio increased (Investigations) | 14 (18) | 5 (6)
Neutrophil count decreased (Investigations) | 40 (167) | 12 (28)
Platelet count decreased (Investigations) | 54 (253) | 28 (76)
Weight decreased (Investigations) | 13 (21) | 3 (4)
Weight increased (Investigations) | 14 (18) | 2 (6)
White blood cell count decreased (Investigations) | 34 (130) | 19 (27)
Decreased appetite (Metabolism and nutrition disorders) | 46 (58) | 20 (22)
Dehydration (Metabolism and nutrition disorders) | 14 (17) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 38 (64) | 13 (18)
Hyperkalaemia (Metabolism and nutrition disorders) | 24 (51) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 24 (33) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 33 (70) | 7 (11)
Hypocalcaemia (Metabolism and nutrition disorders) | 49 (113) | 6 (14)
Hypokalaemia (Metabolism and nutrition disorders) | 72 (194) | 33 (48)
Hypomagnesaemia (Metabolism and nutrition disorders) | 41 (71) | 12 (15)
Hyponatraemia (Metabolism and nutrition disorders) | 32 (78) | 6 (7)
Hypophosphataemia (Metabolism and nutrition disorders) | 43 (77) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 32 (49) | 6 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 33 (37) | 13 (13)
Bone pain (Musculoskeletal and connective tissue disorders) | 14 (16) | 3 (4)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 19 (22) | 1 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 14 (16) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 36 (48) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 37 (45) | 8 (11)
Dizziness (Nervous system disorders) | 48 (66) | 2 (2)
Dysgeusia (Nervous system disorders) | 22 (26) | 4 (4)
Headache (Nervous system disorders) | 62 (89) | 16 (18)
Paraesthesia (Nervous system disorders) | 22 (27) | 0 (0)
Anxiety (Psychiatric disorders) | 19 (22) | 1 (1)
Depression (Psychiatric disorders) | 13 (16) | 7 (7)
Insomnia (Psychiatric disorders) | 42 (46) | 6 (6)
Haematuria (Renal and urinary disorders) | 19 (21) | 5 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 72 (102) | 11 (13)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 52 (70) | 7 (8)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 16 (19) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 42 (51) | 8 (8)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 18 (21) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 21 (24) | 8 (8)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 17 (18) | 2 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 18 (23) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 15 (19) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 14 (18) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 25 (30) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 37 (55) | 10 (10)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 11 (16) | 6 (6)
Hypertension (Vascular disorders) | 35 (77) | 10 (10)
Hypotension (Vascular disorders) | 40 (47) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2020-12-07): https://cdn.clinicaltrials.gov/large-docs/39/NCT02421939/Prot_002.pdf
  • Statistical Analysis Plan (2022-05-31): https://cdn.clinicaltrials.gov/large-docs/39/NCT02421939/SAP_003.pdf